CLINICAL TRIAL: NCT02358772
Title: Comparison of Pre-hospital and In-hospital Iv-tPA Stroke Treatment
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Heinrich J Audebert, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: STEMO_Outcome Analysis
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Stroke
Keywords: stroke; thrombolysis; STEMO
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-hospital thrombolysis: Patients with acute ischemic stroke who are cared in a specialized STroke Emergency MObile (STEMO) before admission to the Hospital and receive thrombolytic therapy (either in STEMO or in Hospital).
  Interventions: Other: thrombolysis in a pre-hospital setting (STEMO concept)
- In-hospital thrombolysis: Patients with acute ischemic stroke who receive thrombolytic therapy after admission to an University Hospital.

INTERVENTIONS:
Other: thrombolysis in a pre-hospital setting (STEMO concept)
  Groups: Pre-hospital thrombolysis

SUMMARY:
This is a comparison of clinical outcomes between a pre-hospital and an in-hospital thrombolysis patient registry.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke diagnosis with thrombolytic treatment
* Admission via EMS
* Known premorbid status of need of assistance
* NIHSS before treatment available
* Time of onset (or last well seen) between 4:00am and 10:30pm

Exclusion Criteria:

* Unknown time of onset
* In-hospital thrombolysis despite decision against treatment because of contraindications in STEMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients with thrombolytic treatment
Sampling Method: Non-Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2011-02; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score | three months after event
  dichotomized mRS 0-1 and 2-6 in patients who lived at home without assistance prior to the index stroke.

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) score | three months after event
  dichotomized mRS 1-3 and 4-6
modified Rankin Scale (mRS) score | three months after event
  mortality (mRS=6)
modified Rankin Scale (mRS) score | three months after event
  ordinal analysis across whole mRS range

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich J Audebert, MD, Principal Investigator — Center for Stroke Research Berlin, Charité Universitätsmedizin Berlin
Locations (1):
- Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Ebinger M, Winter B, Wendt M, Weber JE, Waldschmidt C, Rozanski M, Kunz A, Koch P, Kellner PA, Gierhake D, Villringer K, Fiebach JB, Grittner U, Hartmann A, Mackert BM, Endres M, Audebert HJ; STEMO Consortium. Effect of the use of ambulance-based thrombolysis on time to thrombolysis in acute ischemic stroke: a randomized clinical trial. JAMA. 2014 Apr 23-30;311(16):1622-31. doi: 10.1001/jama.2014.2850. PMID 24756512
- [Background] Kunz A, Ebinger M, Geisler F, Rozanski M, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Fiebach JB, Villringer K, Erdur H, Scheitz JF, Tutuncu S, Bollweg K, Grittner U, Kaczmarek S, Endres M, Nolte CH, Audebert HJ. Functional outcomes of pre-hospital thrombolysis in a mobile stroke treatment unit compared with conventional care: an observational registry study. Lancet Neurol. 2016 Sep;15(10):1035-43. doi: 10.1016/S1474-4422(16)30129-6. Epub 2016 Jul 16. PMID 27430529
- [Derived] Nolte CH, Ebinger M, Scheitz JF, Kunz A, Erdur H, Geisler F, Braemswig TB, Rozanski M, Weber JE, Wendt M, Zieschang K, Fiebach JB, Villringer K, Grittner U, Kaczmarek S, Endres M, Audebert HJ. Effects of Prehospital Thrombolysis in Stroke Patients With Prestroke Dependency. Stroke. 2018 Mar;49(3):646-651. doi: 10.1161/STROKEAHA.117.019060. Epub 2018 Feb 19. PMID 29459395